CLINICAL TRIAL: NCT04456348
Title: Association Between Gait Features Assessed by Artificial Intelligent System and Cognitive Function Decline in the Patients of Silent Cerebrovascular Disease: A Multicenter Prospective Cohort Study
Brief Title: Association Between Gait Assessed by Intelligent System and Cognitive Function in Silent Cerebrovascular Disease
Acronym: ACCURATE-2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: The Affiliated Hospital Of Guizhou Medical University (Other); Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018YFC1312900-01
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2019-11

CONDITIONS: Silent Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- positive: Subjects have gait disorder according to intelligent gait assessment at baseline.
  Interventions: Other: there is no intervention
- negative: Subjects don't have gait disorder according to intelligent gait assessment at baseline.
  Interventions: Other: there is no intervention

INTERVENTIONS:
Other: there is no intervention — There is no intervention

SUMMARY:
This study is a multi-center prospective cohort study. We will continuously recruit subjects with silent cerebrovascular disease aged 60 to 85 years from Shanghai and Guizhou. Data including demographic characteristics, medical history, other concomitant diseases, neurological function assessments, laboratory examinations, imaging examinations, and other clinical data and health economics survey responses will be collected from all subjects.

At baseline, all subjects will undergo gait assessment using the intelligent system and cognitive function scale assessment by clinicians. According to the intelligent gait results, the subjects will be divided into normal and abnormal gait groups. All subjects will be observed naturally for 1 year, and all medical behaviors will be recorded. All subjects will be interviewed by telephone for the occurrence of vascular events and changes in medical behaviors at half a year after enrollment and followed up at 1 year after enrollment, including gait evaluation using the intelligent system and cognitive function scale evaluation by clinicians. During the follow-up period, patients can visit the hospital for follow-up at any time when their condition changes.

DETAILED DESCRIPTION:
The neurological function of all subjects was assessed based on the following tests under the guidance of a physician. The timed up-and-go test was used to evaluate the subjects' gait function, requiring them to stand up from their seat and walk straight forward for 3 meters, turn around, walk straight back to the chair, and then sit down again. Using simple cognitive evaluation (Mini-Cognitive Assessment) screening of the subjects' memory and executive function, the participants will first be asked to remember three unrelated words and immediately repeat the three words; they will then be asked to draw a clock marked with the numbers and pointers, and eventually recall the three words. The verbal function of the subjects will be assessed using the verbal retelling items in the MMSE and Montreal Cognitive Assessment, asking the subjects to clearly repeat "44 stone lions," "I only know Zhang Liang came to help today," and "the cat always hid under the sofa when the dog was in the room." Through the camera image data record, the intelligent system uses the built-in intelligent algorithm for intelligent video gait recognition and neural networks based on depth interpretation automation and automatic access to the subjects' gait characteristics (stand-up time, turnaround time, stride length, step velocity, stride length, step width, etc.), language features (pronunciation, intonation, word order, language accuracy, language fluency, etc.), and clock features.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 60 and 85 years.
2. Diagnosed with silent cerebrovascular disease/silent stroke, which is consistent with the 2016 statement issued by the American Heart Association (AHA) and American Stroke Association (ASA):

   1. No previous clear history of stroke and no clinical symptoms or mild clinical symptoms that fail to attract clinical attention;
   2. Cranial MRI showing at least one of the following within 5 years: lacunar infarct of vascular origin; white matter hyperintensity of vascular origin; cerebral microbleeds;
3. Consciousness and ability to complete cognitive assessment
4. Ability to stand and walk independently and complete gait assessment without assistance from others.
5. Ability to sign the informed consent.

Exclusion Criteria:

1. Intracranial lesions that have been clearly diagnosed as demyelination disease, white matter dystrophy, intracranial space-occupying lesions, or autoimmune encephalitis.
2. Gait disorder that has been diagnosed as Parkinson's disease, normal cranial hydrocephalus, an otogenic disease, subacute combined degeneration, peripheral neuropathy, osteoarthritis, or lumbar disease.
3. Cognitive disorders that have been diagnosed, such as Alzheimer's disease, frontotemporal dementia, Lewy body dementia, etc.
4. Severe neurological diseases such as previous cerebral trauma, epilepsy, and myelopathy, etc.
5. Severe cardiovascular complications and intolerance to the assessment
6. Severe visual or hearing impairment, aphasia, cognitive disorder, gait disorder, etc., that results in the inability to cooperate for cognitive and gait assessment
7. Refusal to participate in the study
8. Other anomalies that could not be included in the exclusion criteria, but are considered inappropriate to be included in this study.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: with silent cerebrovascular disease patient aged 60 to 85 in Shanghai and Guizhou
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive assessment scale score(MMSE) | 1 year
  It will be assessed by the Mini-Mental state examination (MMSE), which is scored 0-30.

SECONDARY OUTCOMES:
Change in cognitive assessment scale score(MoCA) | 1 year
  It will be assessed by the Montreal cognitive assessment (MoCA), which is scored 0-30.
the prevalence of gait disorders | baseline
  the prevalence of gait disorders, according to the intelligent assessment
the prevalence of cognitive disorder | baseline
  the prevalence of cognitive disorder, according to the MMSE
the incidence of vascular events | 1 year
  the incidence of vascular events, including Cardiovascular and cerebrovascular events
the incidence of fall incidence | 1 year
  the incidence of fall incidence

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ding, MD, Study Director — Shanghai Zhongshan Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poels MM, Steyerberg EW, Wieberdink RG, Hofman A, Koudstaal PJ, Ikram MA, Breteler MM. Assessment of cerebral small vessel disease predicts individual stroke risk. J Neurol Neurosurg Psychiatry. 2012 Dec;83(12):1174-9. doi: 10.1136/jnnp-2012-302381. Epub 2012 Aug 23. PMID 22917672
- [Background] Kim BJ, Lee SH. Prognostic Impact of Cerebral Small Vessel Disease on Stroke Outcome. J Stroke. 2015 May;17(2):101-10. doi: 10.5853/jos.2015.17.2.101. Epub 2015 May 29. PMID 26060797
- [Background] Sachdev PS, Wen W, Christensen H, Jorm AF. White matter hyperintensities are related to physical disability and poor motor function. J Neurol Neurosurg Psychiatry. 2005 Mar;76(3):362-7. doi: 10.1136/jnnp.2004.042945. PMID 15716527
- [Background] Murray ME, Senjem ML, Petersen RC, Hollman JH, Preboske GM, Weigand SD, Knopman DS, Ferman TJ, Dickson DW, Jack CR Jr. Functional impact of white matter hyperintensities in cognitively normal elderly subjects. Arch Neurol. 2010 Nov;67(11):1379-85. doi: 10.1001/archneurol.2010.280. PMID 21060015
- [Background] Wakefield DB, Moscufo N, Guttmann CR, Kuchel GA, Kaplan RF, Pearlson G, Wolfson L. White matter hyperintensities predict functional decline in voiding, mobility, and cognition in older adults. J Am Geriatr Soc. 2010 Feb;58(2):275-81. doi: 10.1111/j.1532-5415.2009.02699.x. Epub 2010 Jan 26. PMID 20374403
- [Background] Debette S, Markus HS. The clinical importance of white matter hyperintensities on brain magnetic resonance imaging: systematic review and meta-analysis. BMJ. 2010 Jul 26;341:c3666. doi: 10.1136/bmj.c3666. PMID 20660506
- [Background] Brickman AM, Provenzano FA, Muraskin J, Manly JJ, Blum S, Apa Z, Stern Y, Brown TR, Luchsinger JA, Mayeux R. Regional white matter hyperintensity volume, not hippocampal atrophy, predicts incident Alzheimer disease in the community. Arch Neurol. 2012 Dec;69(12):1621-7. doi: 10.1001/archneurol.2012.1527. PMID 22945686
- [Background] Maillard P, Carmichael O, Fletcher E, Reed B, Mungas D, DeCarli C. Coevolution of white matter hyperintensities and cognition in the elderly. Neurology. 2012 Jul 31;79(5):442-8. doi: 10.1212/WNL.0b013e3182617136. Epub 2012 Jul 18. PMID 22815562
- [Background] Smith EE, Saposnik G, Biessels GJ, Doubal FN, Fornage M, Gorelick PB, Greenberg SM, Higashida RT, Kasner SE, Seshadri S; American Heart Association Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Functional Genomics and Translational Biology; and Council on Hypertension. Prevention of Stroke in Patients With Silent Cerebrovascular Disease: A Scientific Statement for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2017 Feb;48(2):e44-e71. doi: 10.1161/STR.0000000000000116. Epub 2016 Dec 15. PMID 27980126
- [Background] Feigin VL, Forouzanfar MH, Krishnamurthi R, Mensah GA, Connor M, Bennett DA, Moran AE, Sacco RL, Anderson L, Truelsen T, O'Donnell M, Venketasubramanian N, Barker-Collo S, Lawes CM, Wang W, Shinohara Y, Witt E, Ezzati M, Naghavi M, Murray C; Global Burden of Diseases, Injuries, and Risk Factors Study 2010 (GBD 2010) and the GBD Stroke Experts Group. Global and regional burden of stroke during 1990-2010: findings from the Global Burden of Disease Study 2010. Lancet. 2014 Jan 18;383(9913):245-54. doi: 10.1016/s0140-6736(13)61953-4. PMID 24449944
- [Background] Leary MC, Saver JL. Annual incidence of first silent stroke in the United States: a preliminary estimate. Cerebrovasc Dis. 2003;16(3):280-5. doi: 10.1159/000071128. PMID 12865617
- [Background] Vermeer SE, Hollander M, van Dijk EJ, Hofman A, Koudstaal PJ, Breteler MM; Rotterdam Scan Study. Silent brain infarcts and white matter lesions increase stroke risk in the general population: the Rotterdam Scan Study. Stroke. 2003 May;34(5):1126-9. doi: 10.1161/01.STR.0000068408.82115.D2. Epub 2003 Apr 10. PMID 12690219
- [Background] Kim YJ, Kwon HK, Lee JM, Cho H, Kim HJ, Park HK, Jung NY, San Lee J, Lee J, Jang YK, Kim ST, Lee KH, Choe YS, Kim YJ, Na DL, Seo SW. Gray and white matter changes linking cerebral small vessel disease to gait disturbances. Neurology. 2016 Mar 29;86(13):1199-207. doi: 10.1212/WNL.0000000000002516. Epub 2016 Mar 2. PMID 26935893
- [Background] de Laat KF, van Norden AG, Gons RA, van Oudheusden LJ, van Uden IW, Bloem BR, Zwiers MP, de Leeuw FE. Gait in elderly with cerebral small vessel disease. Stroke. 2010 Aug;41(8):1652-8. doi: 10.1161/STROKEAHA.110.583229. Epub 2010 Jun 24. PMID 20576951
- [Background] Montero-Odasso MM, Sarquis-Adamson Y, Speechley M, Borrie MJ, Hachinski VC, Wells J, Riccio PM, Schapira M, Sejdic E, Camicioli RM, Bartha R, McIlroy WE, Muir-Hunter S. Association of Dual-Task Gait With Incident Dementia in Mild Cognitive Impairment: Results From the Gait and Brain Study. JAMA Neurol. 2017 Jul 1;74(7):857-865. doi: 10.1001/jamaneurol.2017.0643. PMID 28505243
- [Background] Wardlaw JM, Smith EE, Biessels GJ, Cordonnier C, Fazekas F, Frayne R, Lindley RI, O'Brien JT, Barkhof F, Benavente OR, Black SE, Brayne C, Breteler M, Chabriat H, Decarli C, de Leeuw FE, Doubal F, Duering M, Fox NC, Greenberg S, Hachinski V, Kilimann I, Mok V, Oostenbrugge Rv, Pantoni L, Speck O, Stephan BC, Teipel S, Viswanathan A, Werring D, Chen C, Smith C, van Buchem M, Norrving B, Gorelick PB, Dichgans M; STandards for ReportIng Vascular changes on nEuroimaging (STRIVE v1). Neuroimaging standards for research into small vessel disease and its contribution to ageing and neurodegeneration. Lancet Neurol. 2013 Aug;12(8):822-38. doi: 10.1016/S1474-4422(13)70124-8. PMID 23867200
- [Result] Vermeer SE, Longstreth WT Jr, Koudstaal PJ. Silent brain infarcts: a systematic review. Lancet Neurol. 2007 Jul;6(7):611-9. doi: 10.1016/S1474-4422(07)70170-9. PMID 17582361
- [Result] Verghese J, Lipton RB, Hall CB, Kuslansky G, Katz MJ, Buschke H. Abnormality of gait as a predictor of non-Alzheimer's dementia. N Engl J Med. 2002 Nov 28;347(22):1761-8. doi: 10.1056/NEJMoa020441. PMID 12456852
- [Result] Dumurgier J, Artaud F, Touraine C, Rouaud O, Tavernier B, Dufouil C, Singh-Manoux A, Tzourio C, Elbaz A. Gait Speed and Decline in Gait Speed as Predictors of Incident Dementia. J Gerontol A Biol Sci Med Sci. 2017 May 1;72(5):655-661. doi: 10.1093/gerona/glw110. PMID 27302701
- [Derived] Tang YM, Fei BN, Li X, Zhao J, Zhang W, Qin GY, Hu M, Ding J, Wang X. Association between gait features assessed by artificial intelligent system and cognitive function decline in patients with silent cerebrovascular disease: study protocol of a multicenter prospective cohort study (ACCURATE-2). BMC Neurol. 2022 Jun 30;22(1):240. doi: 10.1186/s12883-022-02767-2. PMID 35773649